CLINICAL TRIAL: NCT01840826
Title: Reducing Hospital Readmission Among Medical Patients With Depressive Symptoms
Brief Title: Reducing Hospital Readmissions in Patients With Depressive Symptoms
Acronym: RED-D
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Brian Jack, Professor and Chair, Boston Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: H-31632; 1R01HS019700 (AHRQ)
Record Dates: First submitted 2013-04-18; First posted 2013-04-26 (Estimated); Last update posted 2018-03-07 (Actual); Status verified 2018-03

CONDITIONS: Depression
Keywords: Rehospitalization; Reutilization; Depressive Symptoms; Pharmacotherapy; Cognitive Therapy; Self-help; Complementary Therapies
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RED-D Care Management (Experimental): Patients randomized to receive the Intervention work with a RED-D Care Manager post-discharge. The Care Manager meets with the patient in the hospital, prior to discharge, and post-discharge via weekly phone calls. Patients have access to a range of treatment options, overseen by the Care Manager, including: (1) medication; (2) cognitive behavioral therapy (CBT); (3) complementary and alternative medicine (CAM) information and referral; (4) Self-help, such as reading a book, making a change in diet and/or exercise in order to improve mood; (5) active surveillance; and (6) any combination of 1, 2, 3, 4 & 5.
  Interventions: Other: RED-D Care Management
- RED and Behavioral Health Referral (No Intervention): Patients randomized to the "control" group will receive the regular RED intervention, including a follow-up phone call two days post-discharge from the hospital to review and confirm medications, and a referral to behavioral health.

INTERVENTIONS:
Other: RED-D Care Management — The Case Management intervention will continue for 12 weeks post-discharge (from the index admission).
  Arms: RED-D Care Management

SUMMARY:
Project Re-Engineered Discharge (Project RED) has previously demonstrated that patients who received the RED were 30% less likely than patients receiving usual care to access inpatient or emergency services within 30 days of discharge. In this project, the investigators add a new dimension to RED by integrating screening, referral and treatment for depression into the original RED intervention and determining if this enhanced intervention increases the effectiveness of RED in preventing readmissions and controlling costs in the 180 days after discharge for patients with signs of depression.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age
* Admitted to any Boston Medical Center inpatient service or for observation
* Screen positive for depressive symptoms (Patient Health Questionnaire - 2 >/= 3)
* Speaks English with health care providers
* Has access to a telephone
* Live in the Boston area and don't plan on leaving the Boston area for more than 2 weeks in the next 6 months
* Screen positive for depressive symptoms (PHQ -9 >/= 10)

Exclusion Criteria:

* Has plans for inpatient rehabilitation, nursing home, or other institutional settings after discharge.
* Suicidal precautions
* Sickle Cell Crisis (SCC)
* Alcohol and/or drug dependence
* Diagnosis of Bipolar Disorder, Schizophrenia or other Psychotic Disorder
* In police custody

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 709 (Actual)
Dates: Start 2013-02 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
All-cause readmission rates | 30 days and 90 days post-discharge from hospital at index admission
  The primary hypothesis is to test whether the RED intervention plus the collaborative-care approach for depression (RED-D) will reduce the all-cause 30 and 90 day hospital readmission rates for patients who screen positive for depressive symptoms
All-cause reutilization rates | 30 & 90 days post discharge from index hospitalization
  The primary hypothesis is to test whether the RED intervention plus the collaborative-care approach for depression (RED-D) will reduce the all-cause 30 and 90 day hospital utilization rates for patients who screen positive for depressive symptoms

SECONDARY OUTCOMES:
cost-saving | 90 & 180 after discharge from index hospitalization
  The economic analysis will investigate whether the two interventions are cost saving and whether the RED-D intervention is more cost saving than the RED intervention alone. The principal source of the savings is likely to be from reduced rehospitalizations within the 90 days of study follow-up. Hospital administrative records and insurance company data will be used to gather cost data. Additional costs of the two interventions will be estimated by costing staff time and other resources used. Cost-savings will be estimated by t-test comparisons of the mean costs for the groups; given randomization of patient assignment these will provide unbiased estimates.
Mental Health Related Quality of Life | 30 days and 90 days after discharge from index admission
  The impact of the RED-D Collaborative Care Intervention mental health related quality of life will be ascertained using the Quality of Life Enjoyment and Satisfaction Questionnaire (Q-LES-Q) and Work and Social Adjustment Scale (WSAS) . The investigators will test whether collaborative care for depression can produce a clinically meaningful improvement in mental health related quality of life compared to those patients receiving either usual care or the RED discharge alone.

CONTACTS AND LOCATIONS:
Overall Officials: Brian W Jack, MD, Principal Investigator — Boston University
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mitchell SE, Paasche-Orlow MK, Forsythe SR, Chetty VK, O'Donnell JK, Greenwald JL, Culpepper L, Jack BW. Post-discharge hospital utilization among adult medical inpatients with depressive symptoms. J Hosp Med. 2010 Sep;5(7):378-84. doi: 10.1002/jhm.673. PMID 20577971
- [Background] Jack B, Greenwald J, Forsythe S, O'Donnell J, Johnson A, Schipelliti L, Goodwin M, Burniske GM, Hesko C, Paasche-Orlow M, Manasseh C, Anthony D, Martin S, Hollister L, Jack M, Jhaveri V, Casey K, Chetty VK. Developing the Tools to Administer a Comprehensive Hospital Discharge Program: The ReEngineered Discharge (RED) Program. In: Henriksen K, Battles JB, Keyes MA, Grady ML, editors. Advances in Patient Safety: New Directions and Alternative Approaches (Vol. 3: Performance and Tools). Rockville (MD): Agency for Healthcare Research and Quality (US); 2008 Aug. Available from http://www.ncbi.nlm.nih.gov/books/NBK43688/ PMID 21249944
- [Background] Anthony D, Chetty VK, Kartha A, McKenna K, DePaoli MR, Jack B. Re-engineering the Hospital Discharge: An Example of a Multifaceted Process Evaluation. In: Henriksen K, Battles JB, Marks ES, Lewin DI, editors. Advances in Patient Safety: From Research to Implementation (Volume 2: Concepts and Methodology). Rockville (MD): Agency for Healthcare Research and Quality (US); 2005 Feb. Available from http://www.ncbi.nlm.nih.gov/books/NBK20484/ PMID 21249814
- [Background] Clancy CM. Reengineering hospital discharge: a protocol to improve patient safety, reduce costs, and boost patient satisfaction. Am J Med Qual. 2009 Jul-Aug;24(4):344-6. doi: 10.1177/1062860609338131. Epub 2009 Jun 5. No abstract available. PMID 19502567
- [Derived] Mitchell SE, Reichert M, Howard JM, Krizman K, Bragg A, Huffaker M, Parker K, Cawley M, Roberts HW, Sung Y, Brown J, Culpepper L, Cabral HJ, Jack BW. Reducing Readmission of Hospitalized Patients With Depressive Symptoms: A Randomized Trial. Ann Fam Med. 2022 May-Jun;20(3):246-254. doi: 10.1370/afm.2801. PMID 35606137
- See also: Project RED Website Homepage — http://www.bu.edu/fammed/projectred/index.html